CLINICAL TRIAL: NCT00843635
Title: Pilot Study of Phosphodiesterase-5 Inhibitor Tadalafil (Cialis) as an Immunomodulator in Patients With Oral Cavity and Oropharyngeal Squamous Cell Carcinoma.
Brief Title: Tadalafil in Treating Patients Undergoing Surgery for Cancer of the Oral Cavity or Oropharynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donald T. Weed (Other)
Responsible Party: Sponsor-Investigator, Donald T. Weed, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070918; SCCC-2008006 (Other: UM/Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A - Tadalafil 10mg (Experimental): Patients will receive 10mg/day Tadalafil orally on days 1 - 20 in the absence of unacceptable toxicity.
  Interventions: Drug: Tadalafil
- Arm B - Tadalafil 20mg (Experimental): Patients will receive 20mg/day Tadalafil orally on days 1 - 20 in the absence of unacceptable toxicity.
  Interventions: Drug: Tadalafil
- Arm C - Placebo (Placebo Comparator): Patients receive oral placebo once daily on days 1-20 in the absence of unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tadalafil — Given orally
  Other Names: Cialis
  Arms: Arm A - Tadalafil 10mg; Arm B - Tadalafil 20mg
Other: Placebo — Given orally
  Arms: Arm C - Placebo

SUMMARY:
RATIONALE: Biological therapies, such as tadalafil, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This randomized clinical trial is studying how well tadalafil works in treating patients who are undergoing surgery for cancer of the oral cavity or oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze the phenotype and the function of the tumor-induced suppressive network associated with squamous cell carcinoma (SCC) of the head and neck in patients with SCC of the oral cavity or oropharynx treated with tadalafil followed by definitive surgical resection.
* To analyze the immune response before and after treatment with tadalafil to determine whether or not tadalafil treatment modulates in these patients.
* To compare two doses of tadalafil to determine whether there are measurable differences in immune response in these patients.
* To analyze treatment-related side effects of tadalafil at each of the two doses tested in these patients.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral tadalafil once daily on days 1-20 in the absence of unacceptable toxicity.
* Arm II: Patients receive oral tadalafil (at a higher dose than in arm I) once daily on days 1-20 in the absence of unacceptable toxicity.
* Arm III: Patients receive oral placebo once daily on days 1-20 in the absence of unacceptable toxicity.

All patients undergo scheduled definitive surgical resection on day 23.

Patients undergo blood sample collection at baseline, on day 20, and at 6 weeks after surgical resection for correlative laboratory studies. Patients also undergo tumor tissue sample collection at baseline and at the time of surgical resection. Samples are analyzed for immunological markers by Fluorescence-activated cell sorting (FACS) and Immunohistochemistry (IHC).

After completion of study treatment, patients are followed periodically for at least 3 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with surgically resectable oral cavity SCC, all subsites, T1 - T4, N0 - N3
* Patients with surgically resectable oropharyngeal SCC, all subsites, T1 - T2, N0 - N1
* Patients with surgically resectable T4 oropharyngeal SCC, all subsites, N0 - N3
* Patients must be 18 years old or older

EXCLUSION CRITERIA:

* Patients with previous surgical resection, radiation, or chemotherapy will be excluded to rule out possible effects of local tissue changes secondary to previous treatment
* Patients with surgically unresectable disease at primary site or regional lymph nodes
* Patients with T1 - T2 SCC oropharynx, N2 - N3
* Patients with T3 SCC oropharynx , N0 - N3
* Any patient for whom non-surgical therapy is recommended as treatment of choice after multidisciplinary treatment evaluation
* Patients with an altered mental status or not capacitated for their medical decision making
* Patients with severe or unstable cardiac or cerebrovascular disease are excluded

  * myocardial infarction within the last 90 days
  * unstable angina or angina occurring during sexual intercourse
  * New York Heart Association Class 2 or greater heart failure in the last 6 months
  * uncontrolled arrhythmias
  * hypotension (<90/50 mm Hg), or uncontrolled hypertension (>170/100 mm Hg)
  * stroke within the last 6 months
  * Left ventricle outflow obstruction.
* Pregnant and nursing mothers will not be enrolled given unknown effects to offspring
* Concurrent nitrate, alpha-blocker, or cytochrome P-450 inhibitor use
* Renal Insufficiency defined as creatinine clearance less than 51.
* Creatinine clearance will be determined by the following Cockcroft-Gault Equation: (140-age) * (Wt in kg) * (0.85 if female) / (72 * Cr)
* Patients with hepatic insufficiency.
* Patients currently taking a Phosphodiesterase (PDE) inhibitors for erectile dysfunction
* Patients who are immunocompromised, for reasons not directly related to patients malignancy
* Patients with significant alcohol or drug abuse
* Patients with unilateral blindness, hereditary retinal disorders, or increased risk of blindness
* Patients with unilateral deafness, history of hearing loss, hearing aid dependence, or clinically evident hearing loss

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald T. Weed, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Weed DT, Vella JL, Reis IM, De la Fuente AC, Gomez C, Sargi Z, Nazarian R, Califano J, Borrello I, Serafini P. Tadalafil reduces myeloid-derived suppressor cells and regulatory T cells and promotes tumor immunity in patients with head and neck squamous cell carcinoma. Clin Cancer Res. 2015 Jan 1;21(1):39-48. doi: 10.1158/1078-0432.CCR-14-1711. Epub 2014 Oct 15. PMID 25320361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Started | 15 | 15 | 5
Completed | 13 | 13 | 5
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Race/ethnicity reported for 34 of the 35 participants, specifically for 14 of the 15 participants in Arm B - Tadalafil 20mg.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo | Total
Number analyzed (Participants) | 15 | 15 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.5) | 59 (13.9) | 66.8 (4.3) | 60.3 (11.6)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [39 to 76] | 54 [39 to 81] | 67 [60 to 72] | 63 [39 to 81]
Age, Customized [Number; unit: participants]
  < 50 years of age | 2 | 6 | 0 | 8
  50 to 59 years of age | 5 | 2 | 0 | 7
  60 to 69 years of age | 5 | 3 | 4 | 12
  70+ years of age | 3 | 4 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 12 | 11 | 4 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  White, Non-Hispanic | 12 | 8 | 3 | 23
  Hispanic | 3 | 5 | 2 | 10
  South Asian | 0 | 1 | 0 | 1
  Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 35
Alcohol Use [Number; unit: participants]
  Never | 2 | 2 | 1 | 5
  Current Use | 11 | 8 | 4 | 23
  Past Use | 2 | 5 | 0 | 7
Tobacco Use [Number; unit: participants]
  Current | 9 | 9 | 0 | 18
  Quit < 20 years ago | 3 | 1 | 4 | 8
  Quit > 20 years ago | 0 | 3 | 0 | 3
  Never | 3 | 2 | 1 | 6
Type of Tobacco Use [Number; unit: participants]
  Never | 3 | 2 | 1 | 6
  Cigarettes | 12 | 11 | 4 | 27
  Cigar/Pipe | 0 | 1 | 0 | 1
  Snuff/Chew/Smokeless | 0 | 1 | 0 | 1
Site [Number; unit: participants]
  Oral Cavity | 13 | 14 | 4 | 31
  Oro Pharynx | 2 | 1 | 1 | 4
Tumor size (cm) Mean [Mean (Standard Deviation); unit: cm] | 3.7 (1.8) | 2.4 (1.3) | 3.5 (1.9) | 3.1 (1.7)
Tumor Size (cm) Median [Median (Inter-Quartile Range); unit: cm] | 3 [2 to 8.5] | 2.1 [0.5 to 5.5] | 4 [0.6 to 5.5] | 3 [0.5 to 8.5]
T-Stage [Number; unit: participants] — Number of participants on each arm grouped by the size and/or extent (reach) of the primary tumor (T) at Baseline: T1, T2, T3 and T4.
  Numbers after the T (such as T1, T2, T3, and T4) might describe the tumor size and/or amount of spread into nearby structures. The higher the T number, the larger the tumor and/or the more it has grown into nearby tissues.
  participants
    T1 | 1 | 7 | 1 | 9
    T2 | 9 | 4 | 2 | 15
    T3 | 1 | 0 | 1 | 2
    T4 | 4 | 4 | 1 | 9
N Stage - Regional Lymph Nodes [Number; unit: participants] — Number of participants on each arm grouped by whether or not the cancer has reached nearby lymph nodes at Baseline:
  * N0 - No regional lymph node involvement (no cancer found in the lymph nodes)
  * N1 - N3 - Involvement of regional lymph nodes (number and/or extent of spread)
  participants
    N0 | 7 | 9 | 4 | 20
    N1 | 2 | 1 | 1 | 4
    N2b | 4 | 3 | 0 | 7
    N2c | 1 | 2 | 0 | 3
    N3 | 1 | 0 | 0 | 1
Positive for Human Papillomavirus (HPV+) [Number; unit: participants]
  Yes | 3 | 1 | 0 | 4
  No | 12 | 14 | 5 | 31
Pre-Operative Treatment [Number; unit: participants]
  No | 10 | 13 | 3 | 26
  Yes | 5 | 2 | 2 | 9
Pre-Operative Treatment, Details [Number; unit: participants]
  No | 10 | 13 | 3 | 26
  Chemo + Radiation | 1 | 1 | 2 | 4
  Radiation only | 4 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Ratio of MDSC Concentration in the Blood
Description: Ratio of the number of Myeloid Derived Suppressor Cells (MDSC) in the Blood, per treatment group, from Baseline to End of Treatment at Time of Surgery.
Time Frame: Baseline, End of Treatment at time of Surgery
Measure: Median (Inter-Quartile Range); unit: ratio from baseline
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Number analyzed (Participants) | 13 | 13 | 5
ratio from baseline | 0.7680 [0.6440 to 1.010] | 0.7919 [0.4344 to 1.115] | 0.9876 [0.8478 to 1.026]

2. Primary Outcome: Ratio of T-reg Cell Concentration in the Blood
Description: Ratio of the number of regulatory T cells in the blood, per treatment group, from Baseline to End of Treatment at Time of Surgery..
Time Frame: Baseline, End of Treatment at Time of Surgery
Measure: Median (Inter-Quartile Range); unit: ratio from baseline
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Number analyzed (Participants) | 13 | 13 | 5
ratio from baseline | 0.7776 [0.5751 to 0.8869] | 0.6789 [0.5234 to 1.033] | 0.8421 [0.5255 to 0.9142]

3. Primary Outcome: Ratio of Tumor-specific T-cell Concentration in the Blood
Description: Ratio of the number of tumor specific T cells in the blood, per treatment group, from Baseline to End of Treatment at Time of Surgery.
Time Frame: Baseline, End of Treatment at Time of Surgery
Population: Data for 31 patients were analyzed.
Measure: Median (Inter-Quartile Range); unit: ratio from baseline
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Number analyzed (Participants) | 12 | 10 | 3
ratio from baseline | 1.7401 [1.1478 to 2.7495] | 1.9020 [1.0413 to 6.1008] | 1.0933 [0.7884 to 1.2466]

4. Secondary Outcome: Optimal Dosing Schedule for Tadalafil
Time Frame: Baseline, End of Treatment at Time of Surgery.
Population: Optimal dosing schedule of Tadalafil not determined due to no proven superiority of one dosing arm over the other.
Groups:
- Arm A (Tadalafil 10mg) + Arm B (Tadalafil 20mg): All participants enrolled to the two dosing arms, Arm A (Tadalafil 10 mg) and Arm B (Tadalafil 20 mg).
Arm/Group | Arm A (Tadalafil 10mg) + Arm B (Tadalafil 20mg)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Assessment of Treatment-related Side Effects. Number of participants experiencing adverse events
Time Frame: From Day 1 to Day 20
Measure: Number; unit: participants
Groups:
- Arm A - 10mg: Patients will receive 10mg/day Tadalafil orally on days 1 - 20 in the absence of unacceptable toxicity.
Arm/Group | Arm A - 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Number analyzed (Participants) | 15 | 15 | 5
participants | 4 | 10 | 3

ADVERSE EVENTS:
Arm/Group | Arm A - Tadalafil 10mg | Arm B - Tadalafil 20mg | Arm C - Placebo
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/15 | 0/5
Other Adverse Events (participants affected / at risk) | 3/15 | 8/15 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Tadalafil 10mg (N=15) | Arm B - Tadalafil 20mg (N=15) | Arm C - Placebo (N=5)
Back Pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia - Grade 3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Tadalafil 10mg (N=15) | Arm B - Tadalafil 20mg (N=15) | Arm C - Placebo (N=5)
Back Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache - Grade 2 (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain - Grade 2 (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity - Grade 2 (General disorders) | 0 (0) | 1 (2) | 0 (0)
Back Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough - Grade 1 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ear Nose Throat Examination abnormal (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Headache - Grade 1 (General disorders) | 0 (0) | 1 (2) | 2 (2)
Neck Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Pain in Extremity - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sexual - Grade 1 (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Race/Ethnicity baseline characteristics reported for 34 of 35 patients enrolled. Data analyzed for outcome measure for the 31 participants who completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes